CLINICAL TRIAL: NCT05736315
Title: Phase II Randomized, Double Blind Study of Probiotics in Patients With Cervical Cancer in Clinical Stages IIB Undergoing Concurrent Chemotherapy and Radiation Therapy
Brief Title: Use of a Fermented Dairy Beverage in Cervical Cancer Patients Undergoing Concurrent Chemoradiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: Yakult Honsha Co., LTD (Industry); Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other); Instituto Nacional de Perinatologia (Other Government)
Responsible Party: Principal Investigator, Dr. Lucely Cetina Pérez, Principal investigator, National Institute of Cancerología
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 008/043/ICI
Record Dates: First submitted 2023-01-31; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Cervical Cancer, Stage IIB
Keywords: Cervical cancer; Probiotics; Toxicity; Inflammation; Quality of Life
MeSH Terms: conditions — Uterine Cervical Neoplasms; Inflammation | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented dairy beverage (Experimental): Concumption of 3 servings of the fermented dairy beverage a day, during oncological treatment.
  Interventions: Other: Placebo dairy beverage
- Placebo (Placebo Comparator): Consumption of 3 servings of the placebo dairy beverage a day, during oncological treatment.
  Interventions: Other: Placebo dairy beverage

INTERVENTIONS:
Other: Placebo dairy beverage — Placebo dairy beverage (placebo) is a sweetened dairy beverage.
  Other Names: Probiotic

SUMMARY:
Many cancer survivors have increased risk of intestinal damage, affecting the quality of life of patients. The role of intestinal microbiota on the development of gastrointestinal toxicity and radiation enteritis has been described in cervical cancer patients that received pelvic RT. In this project we investigated the effect that a fermented dairy beverage (Yakult) may have in the modulation of inflammation and consequently of gastrointestinal toxicity in locally advanced cervical cancer (LACC) patients treated with concomitant chemo-radiotherapy (CRT).

DETAILED DESCRIPTION:
Globally, many cancer survivors have undergone radiotherapy (RT) to pelvic tumors, this confers an increased risk of intestinal damage, affecting the quality of life of patients. The role of intestinal microbiota on the development of gastrointestinal toxicity and radiation enteritis has been described in cervical cancer patients that received pelvic RT. In this project we investigated the effect that a fermented dairy beverage (Yakult) may have in the modulation of inflammation and consequently of gastrointestinal toxicity in locally advanced cervical cancer (LACC) patients treated with concomitant chemo-radiotherapy (CRT).

In Mexico, the incidence of cervical cancer is 23 cases in 100,000 women (2015, Secretaría de Salud). In the Mexican National Cancer Institute (Instituto Nacional de Cancerología; INCan), 80% of patients arrive at locally advanced stages (IB2-IVA), the standard treatment is based on CRT. Gastrointestinal symptoms experienced by patients that receive pelvic RT define the pelvic radiation disease (PRD). Acute PRD is the result of cell death in the crypt epithelium and an acute inflammatory response in the lamina propria, which results in an insufficient replacement of the villi, rupture and inflammation of the mucosal barrier. Symptoms develop in 60-80% of patients. These include nausea, diarrhea, tenesmus, abdominal pain, urgency, anorexia, bleeding and fatigue; these are dose-limiting symptoms and affect the patients' quality of life.

A recent study analyzed the microbiota of LACC patients and found that patients that develop PRD during treatment with CRT possess a different microbiota to those patients that do not develop severe gastrointestinal toxicity. Evidence points to the critical role that the microbiota and intestinal inflammation play for the development of PRD in LACC patients. Therefore, an optimal intervention that modulates the microbiota is essential. We aimed to investigate the effect that a dairy beverage fermented with the probiotic Lactobacillus casei Shirota may have on intestinal and systemic inflammation, and consequently gastrointestinal symptoms and quality of life in women with LACC, undergoing CRT.

METHODS. This study was a double blind, placebo-controlled trial for Stage IIB cervical cancer patients that underwent CRT. The intervention group consumed of 3 servings of the fermented dairy beverage (Yakult) a day. The control group consumed 3 servings of the placebo beverage (with the same organoleptic qualities of Yakult). Clinical toxicity was analyzed with the Common Toxicity Criteria Version 2. Quality of Life score was measured with the QLQC 30 EORTC questionnaire. Fecal calprotectin was quantified to determine intestinal inflammation. Pro- and anti-inflammatory cytokines were quantified in blood samples to determine systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of cervical cancer staged as IIB.
* Histology: Epidermoid, adenosquamous, and adenocarcinoma
* Without previous treatment
* Measurable disease
* Age between 18 and 70 years
* Functional status of 0-2 (WHO criteria)
* Normal hematological, renal and hepatic function
* Standard chest X-ray
* Informed consent

Exclusion Criteria:

* Patients with small cell carcinoma or other rare histologies (sarcomas, lymphomas)
* Patients with other clinical stages
* Patients with paraaotic nodes less than or equal to 1 cm.
* Patients with non-measurable disease
* Infections or serious diseases that prevent the use of chemotherapy
* Concomitant treatment with another experimental drug
* Pregnancy or lactation
* Mental diseases
* Patients with previously documented hypersensitivity reactions to lactobacilli.
* Diabetic patients or hyperglycemia higher than 145 mg/dL.
* Previous or concomitant malignancy except non-melanoma skin carcinoma
* Social, family or geographical conditions that suggest a poor adherence to the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-04-25 (Actual); Primary Completion 2007-06-25 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Clinical toxicity | Change from baseline up to 3 months after treatment finished
  Toxicity was analyzed with the Common Toxicity Criteria Version 2.
  A grading (severity) scale is provided for each adverse event (AE) term. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4 Life-threatening consequences; urgent intervention indicated.
  Grade 5 Death related to AE.

SECONDARY OUTCOMES:
Health Related Quality of Life | Change from baseline up to 3 months after treatment finished
  It was measured with the EORTC QLQ-C30 V2.
Pro- and anti-inflammatory cytokines | Change from baseline up to 3 months after treatment finished
  Th1, Th2, Th17 and IL-10 citokines were quantified in blood samples to determine systemic inflammation using immune assay ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Lucely Cetina Pérez, MD, PhD, Principal Investigator — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- National Cancer Institute of Mexico, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No